CLINICAL TRIAL: NCT04946838
Title: Transcutaneous Electrical Nerve Stimulation for Labor Pain Control in Combination With Cardiotocography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Centaflow (Industry)
Responsible Party: Principal Investigator, Kenoja Thuvarakan, Principle Investigator, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20210423
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Labor Pain
Keywords: TENS; Labor pain; Childbirth; RCT; Pilot study
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: 2 groups (TENS and sham)
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS (Experimental): TENS with 4/100 Hz in frequency, 200 µs in pulse duration, and intensity individually adjusted.
  Interventions: Device: DS5 electrical stimulator
- Sham-TENS (Sham Comparator): Sham with 100 Hz in frequency, 200 µs in pulse duration, and intensity below 5 mA.
  Interventions: Device: DS5 electrical stimulator

INTERVENTIONS:
Device: DS5 electrical stimulator — TENS

SUMMARY:
Transcutaneous electrical nerve stimulation (TENS) is a non-invasive electro-physical modality used for several pain conditions including labor pain control. Despite several years of research, there is still no agreement within the literature regarding the selection of TENS parameters. It is aimed to investigate TENS1 alternating between 4 to 100 Hz compared to sham-TENS.

The present study aims to evaluate TENS in combination with cardiotocography (CTG).

The combination of TENS with CTG in a feedback-loop has not been reported in any studies before.

DETAILED DESCRIPTION:
Midwives and the study investigator will ask parturients, who are admitted to the labor ward at Region Hospital Herning satisfying the inclusion and exclusion criteria, whether they are interested in attending the experimental session.

The study will be conducted as soon as the subject is admitted at the labor ward. The study will only be conducted during early and active labor and not during the birth of the baby.

The subject in this study includes the package of a parturient and her neonate (after birth) as we also obtain data about the neonate. Hereby, two consent forms will be obtained. As this study is a non-invasive study, it is decided to have at least the consent of one parent.

The investigator will fill out a screening questionnaire about the laboring parturient in cooperation with the subject and the midwife, including screening questions related to inclusion and exclusion criteria before the experimental session starts.

The study will last approximately one hour and will be conducted during laboring circumstances. KT (Kenoja Thuvarakan) will carry out the experiment, and she will be present in the delivery room during the whole session.

The study includes several outcomes, including subjective and semi-objective pain measures. The primary outcome is VAS (0-10 cm scale), while secondary outcomes include PPT and satisfaction questionnaire (only at the end of the study). The subjects will be asked before, and immediately after the experimental exposure about the outcomes (VAS and PPT). The subjects will be exposed to one of the two combinations of TENS stimulation (low-to-high and high alternating frequency), which will be compared to sham-TENS.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Vertex presentation
* Speak, read and understand Danish

Exclusion Criteria:

* Gestational age < 37+0 weeks
* Gestational age > to 41+6 weeks
* High-risk pregnancies (including risk factors: eclampsia, pre-eclampsia, diabetes, gestational diabetes, hypertension (above 140/90), and hypotension (below 90/60), Intrauterine growth restriction (IUGR), polyhydramnious, and oligohydramnious).
* Pre-gestational body mass index (BMI) above 40 kg/m2
* Use of fetal scalp-electrode during the experiment
* Use of pacemakers and other electronic implants
* Severe arrhythmia
* Present musculoskeletal illnesses (including myopathy and arthritis).
* Chronic pain within last 6 months (Pelvic girdle pain (PGP) to a mild degree (VAS 0-6 cm) is accepted in the experiment. Severe degree (VAS 6-10 cm) (e.g. bedridden or difficulty walking) especially within 24 hours before birth is excluded).
* Present/previous neurologic illnesses (including epilepsy, migraine, and sclerosis).
* Present medicated mental disorders (including dementia, personality disorders, bipolar, ADHD, and anxiety).
* Dermatological disorders (including skin allergy, tattoos or scars on the locations of electrodes)
* Use of other long-acting pain relief before the experiment (including Epidural, Morphine less than 16 hours before experiment), Acupuncture, Paracetamol (less than 8 hours before experiment), Cocktail (less than 8 hours before experiment), nitrous oxide (less than one hour before experiment), sterile water injection (less than two hours before experiment).
* Use of TENS 48 hours before the trial
* Drug addiction defined as the use of cannabis, opioids or other drugs.
* Smokers
* Lack of ability to cooperate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-13 (Actual)

PRIMARY OUTCOMES:
Visual Analog scale (VAS) | Baseline, 10 minutes post stimulation, 30 minutes post stimulation
  10-cm pain intensity scale with 0 cm is no pain and 10 cm is unbearable pain. Decreased cm after baseline measurement indicates pain relief.
Pain pressure threshold (PPT) | Baseline, 10 minutes post stimulation, 30 minutes post stimulation
  Pain sensitivity measurement also defined as the minimum pressure needed to evoke a pain response measured in kPa. Increased kPa after baseline measurement indicates pain relief.

SECONDARY OUTCOMES:
Satisfaction of TENS | Right after last measurements of VAS & PPT
  Satisfaction rating on scale from 0 to 10 [0 as 'no satisfaction' and 10 as 'total satisfaction'].
Experienced pain reduction | Right after last measurements of VAS & PPT
  Response to yes or no
Interest in the use of TENS again | Right after last measurements of VAS & PPT
  Response to yes, no, or don't know
Recommend TENS to others | Right after last measurements of VAS & PPT
  Response to yes, no, or don't know

CONTACTS AND LOCATIONS:
Overall Officials: Parisa Gazerani, PhD, Study Director — Aalborg University
Locations (1):
- Region Hospital Gødstrup, Herning, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and individual participant data will be available.
Supporting Information: Study Protocol
Time Frame: The study protocol will also be published after the manuscript publication. Expected to be published after September 2021.